CLINICAL TRIAL: NCT05261412
Title: Varicose Vein Education and Informed coNsent (VVEIN) Study: A Randomised Feasibility Study
Brief Title: Varicose Vein Education and Informed coNsent (VVEIN) Study
Acronym: VVEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: EIDO Healthcare (Other)
Responsible Party: Principal Investigator, Aoife Kiernan, Research Fellow, Royal College of Surgeons, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RoyalCSI1
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Varicose Veins
Keywords: Informed consent; Educational tool; Digital Consent; Telemedicine; Knowledge recall; Anxiety; Satisfaction
MeSH Terms: conditions — Varicose Veins; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Consent (Control) (Active Comparator): Standard consent (written patient information leaflet (PIL) + verbal discussion with the responsible surgeon) for EVTA followed by signing of consent.
  Interventions: Other: Standard Consent
- Digital health education tool (dHET) (Experimental): dHET for EVTA + verbal discussion with the responsible surgeon followed by signing of consent.
  Interventions: Other: Digital health education tool (dHET)

INTERVENTIONS:
Other: Standard Consent — Participants in the control arm will undergo Standard Consent which will consist of paper PIL provided by EIDO healthcare followed by a verbal discussion (standardized by following a checklist of topics to discuss) with the responsible consultant surgeon and signing of the consent form. The time taken to read the PIL (self-recorded by the patient) will be recorded. The time spent with the responsible surgeon will also be recorded, as will the number of questions asked by the participant.
  Other Names: Paper consent
  Arms: Standard Consent (Control)
Other: Digital health education tool (dHET) — Participants randomized to the intervention dHET will receive the dHET followed by a verbal discussion (as above) and signing of the consent form. The dHET will be delivered on a tablet computer and facilitated by a research assistant who will ensure all technological issues are overcome but will not engage with the participant with regard facilitating better understanding of the content. The digital offering will be interactive; participants will be able to traverse through each section at their own pace with the ability to re-visit sections. It also contains a two-minute narrated animation of the procedure, which can played, rewinded or fast forward. The time spent reading each section of the dHET and time spent watching the animation will be recorded. The time spent with the responsible surgeon will also be recorded, as will the number of questions asked by the participant.
  Other Names: Educational tool; Multimedia consent
  Arms: Digital health education tool (dHET)

SUMMARY:
This is a prospective, single centre, randomised controlled, feasibility study recruiting patients with varicose veins. Patients will be randomised to receive standard (verbal discussion and written information pamphlet) consent or a digital health education tool (dHET). The primary endpoints will be feasibility and practicality of introducing dHET into a busy day surgery practice, secondary endpoints will included knowledge recall of essential information, patient anxiety, patient satisfaction and the time spent in person with the responsible surgeon and number of questions asked prior to signing the consent document.

DETAILED DESCRIPTION:
Varicose Veins (VV) affect one-third of the adult population and chronic venous disease (CVD) has a negative effect on quality of life (QoL), which can be significantly improved by treatment.[1-4] Chronic venous insufficiency (CVI) can be complicated by venous ulceration in over 3% of patients, and chronic treatment with dressings has been estimated to consume 2% of the health budget. Over the last 15 years, minimally invasive endovenous techniques to treat VV have been introduced and are proven to be cost-effective and safe, particularly when performed under a local anaesthetic in an outpatient setting.[5] The American Venous Forum, in 2011, and the National Institute for Health and Care Excellence NICE), in 2013, have recommended endovenous thermal ablation (EVTA) techniques, as the first-line treatments for truncal reflux.[6,7]

As doctors, there is a legal requirement and duty of care to ensure patients are enabled to make an informed decision about their treatment, including discussion of the benefits, risks and alternative treatments. This is reflected in the Health Service Executive (HSE) National Consent Policy and Irish Medical Council 'Guide to Professional Conduct and Ethics'. [8] A patient centered approach to consent has been firmly established in Ireland since 2000, it reinforces that there is a duty to involve patients in decisions about treatments and to engage in a dialogue that offers comprehensible information. This is in keeping with the fundamental ethical principle of autonomy.[8]

Interventions to improve information transfer and comprehension in the consent process [9], such as standard Patient Information Leaflets (PIL) report mixed results. Information leaflets used during the process of consent have been shown to increase patient factual recall and satisfaction with the consent process and are considered best practice. [10-15] However, even well considered PILs, co-designed with patient or client engagement, do not always cover the less common areas of concern or risk which may be material to an individual patient. [9] More rigorous approaches are time and cost intensive, and can adversely impact on the efficiency of healthcare delivery, which limits scalability.

Telemedicine has revolutionised the delivery of care to patients in the modern era of computers, tablets, and smartphones and its use has been rapidly expanded.[16] Digital platforms are a novel tool to potentially improve dialogue and communication between doctors and patients. Patients in general have high satisfaction ratings for telemedicine, but certain patient-groups may be less likely to engage or benefit from it on account of disability, technological illiteracy or access.[16] The use of novel digital technologies can offer a low cost, accessible and tailored solution.

Thus the rationale for this study is to investigate whether it is feasible and acceptable to deliver a digital health education intervention to patients to supplement the consent process.

ELIGIBILITY:
Inclusion Criteria:

* Deemed suitable for EVTA by treating surgeon
* First procedure for superficial venous incompetence
* Full consent
* >18 years
* Proficient in English

Exclusion Criteria:

* Redo or second procedure for superficial venous incompetence (in same or opposite leg)
* Cognitive impairment or unable to consent
* Not meeting inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Eligible participants | Through study completion, an average of 12 months
  Number of eligible participants (meeting inclusion criteria)
Recruitment rate | Through study completion, an average of 12 months
  Number of participants consenting to participate
Retention rate | Through study completion, an average of 12 months
  (Number of patients who consent to participation) minus (number of patients who voluntarily withdraw) divided by (number of subjects who enrol)
Acceptability | Through study completion, an average of 12 months
  Number of patients declining to participate, reasons for declining, number of patients withdrawing consent
Adherence to protocol | Through study completion, an average of 12 months
  Number of patients who adhered to assigned intervention protocol, also includes the proportion of complete data for each outcome measure
Barriers to assigned intervention | Through study completion, an average of 12 months
  Number of patients not randomised due to staffing or time constraints (with reason recorded), technology issues with tablet/dHET/link to knowledge quiz/ internet access
Time | Immediately post intervention
  Time (seconds) taken to complete the assigned intervention (and any delays caused as a result)

SECONDARY OUTCOMES:
Knowledge | Baseline, immediately after intervention, delayed (two week follow up)
  Comprehension test about EVTA using True/False format
Patient Anxiety | Baseline, immediately after intervention, delayed (two week follow up)
  Anxiety measured with short-form State Trait Anxiety Inventory (STAI-6)
Patient Satisfaction | Immediately after intervention and delayed (two week follow up)
  Satisfaction of patients measured with Client satisfaction questionnaire (CSQ-8)
Time spent face to face with surgeon | Post intervention (day of surgery)
  Time spent during verbal discussion of consent with responsible surgeon (measured in seconds)
Questions asked | Post intervention (day of surgery)
  Number of questions asked by patients during consent

CONTACTS AND LOCATIONS:
Overall Officials: Denis Harkin, Study Director — Royal College of Surgeons, Ireland; Aoife Kiernan, Principal Investigator — Royal College of Surgeons, Ireland
Locations (1):
- Bon Secours Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans CJ, Fowkes FG, Ruckley CV, Lee AJ. Prevalence of varicose veins and chronic venous insufficiency in men and women in the general population: Edinburgh Vein Study. J Epidemiol Community Health. 1999 Mar;53(3):149-53. doi: 10.1136/jech.53.3.149. PMID 10396491
- [Background] Smith JJ, Garratt AM, Guest M, Greenhalgh RM, Davies AH. Evaluating and improving health-related quality of life in patients with varicose veins. J Vasc Surg. 1999 Oct;30(4):710-9. doi: 10.1016/s0741-5214(99)70110-2. PMID 10514210
- [Background] MacKenzie RK, Paisley A, Allan PL, Lee AJ, Ruckley CV, Bradbury AW. The effect of long saphenous vein stripping on quality of life. J Vasc Surg. 2002 Jun;35(6):1197-203. doi: 10.1067/mva.2002.121985. PMID 12042731
- [Background] Biemans AA, Kockaert M, Akkersdijk GP, van den Bos RR, de Maeseneer MG, Cuypers P, Stijnen T, Neumann MH, Nijsten T. Comparing endovenous laser ablation, foam sclerotherapy, and conventional surgery for great saphenous varicose veins. J Vasc Surg. 2013 Sep;58(3):727-34.e1. doi: 10.1016/j.jvs.2012.12.074. Epub 2013 Jun 13. PMID 23769603
- [Background] van den Bos R, Arends L, Kockaert M, Neumann M, Nijsten T. Endovenous therapies of lower extremity varicosities: a meta-analysis. J Vasc Surg. 2009 Jan;49(1):230-9. doi: 10.1016/j.jvs.2008.06.030. Epub 2008 Aug 9. PMID 18692348
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] National Clinical Guideline Centre (UK). Varicose Veins in the Legs: The Diagnosis and Management of Varicose Veins. London: National Institute for Health and Care Excellence (NICE); 2013 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK264166/ PMID 25535637
- [Background] Medical Council, The Guide to Professional Conduct and Ethics for Registered Medical Practitioners [2009] para, 9.2
- [Background] Grady C. Enduring and emerging challenges of informed consent. N Engl J Med. 2015 Feb 26;372(9):855-62. doi: 10.1056/NEJMra1411250. PMID 25714163
- [Background] Emanuel EJ, Emanuel LL. Four models of the physician-patient relationship. JAMA. 1992 Apr 22-29;267(16):2221-6. No abstract available. PMID 1556799
- [Background] Gartner FR, Bomhof-Roordink H, Smith IP, Scholl I, Stiggelbout AM, Pieterse AH. The quality of instruments to assess the process of shared decision making: A systematic review. PLoS One. 2018 Feb 15;13(2):e0191747. doi: 10.1371/journal.pone.0191747. eCollection 2018. PMID 29447193
- [Background] Stiggelbout AM, Pieterse AH, De Haes JC. Shared decision making: Concepts, evidence, and practice. Patient Educ Couns. 2015 Oct;98(10):1172-9. doi: 10.1016/j.pec.2015.06.022. Epub 2015 Jul 15. PMID 26215573
- [Background] Couet N, Desroches S, Robitaille H, Vaillancourt H, Leblanc A, Turcotte S, Elwyn G, Legare F. Assessments of the extent to which health-care providers involve patients in decision making: a systematic review of studies using the OPTION instrument. Health Expect. 2015 Aug;18(4):542-61. doi: 10.1111/hex.12054. Epub 2013 Mar 4. PMID 23451939
- [Background] Pascoe GC. Patient satisfaction in primary health care: a literature review and analysis. Eval Program Plann. 1983;6(3-4):185-210. doi: 10.1016/0149-7189(83)90002-2. PMID 10299618
- [Background] Weinstein RS, Lopez AM, Joseph BA, Erps KA, Holcomb M, Barker GP, Krupinski EA. Telemedicine, telehealth, and mobile health applications that work: opportunities and barriers. Am J Med. 2014 Mar;127(3):183-7. doi: 10.1016/j.amjmed.2013.09.032. Epub 2013 Oct 29. PMID 24384059
- [Derived] Kiernan A, Boland F, Moneley D, Doyle F, Harkin DW. Varicose Vein Education and Informed coNsent (VVEIN) study: a randomised controlled pilot feasibility study. Pilot Feasibility Stud. 2023 Jun 22;9(1):104. doi: 10.1186/s40814-023-01336-9. PMID 37349825